CLINICAL TRIAL: NCT01702714
Title: A MULTICENTER, OPEN-LABEL PHASE IB STUDY OF RO5083945 IN COMBINATION WITH CISPLATIN AND GEMCITABINE OR CARBOPLATIN AND PACLITAXEL IN PATIENTS WITH ADVANCED OR RECURRENT NON SMALL CELL LUNG CANCER OF SQUAMOUS HISTOLOGY WHO HAVE NOT RECEIVED PRIOR CHEMOTHERAPY FOR THE METASTATIC DISEASE.
Brief Title: A Study of RO5083945 in Combination With Cisplatin and Gemcitabine or Carboplatin and Paclitaxel in Patients With Advanced or Recurrent Non-Small Cell Lung Cancer of Squamous Histology Who Have Not Received Prior Chemotherapy for The Metastatic Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Project Team decision
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP28577; 2012-003376-39 (EudraCT Number)
Record Dates: First submitted 2012-10-01; First posted 2012-10-08 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — imgatuzumab; Carboplatin; Cisplatin; Gemcitabine; Paclitaxel

ARMS (2):
- RO5083945 + carboplatin + paclitaxel (Experimental)
  Interventions: Drug: RO5083945; Drug: carboplatin; Drug: paclitaxel
- RO5083945 + cisplatin +gemcitabine (Experimental)
  Interventions: Drug: RO5083945; Drug: cisplatin; Drug: gemcitabine

INTERVENTIONS:
Drug: RO5083945 — multiple ascending doses
Drug: carboplatin — up to 6 cycles
  Arms: RO5083945 + carboplatin + paclitaxel
Drug: cisplatin — up to 6 cycles
  Arms: RO5083945 + cisplatin +gemcitabine
Drug: gemcitabine — up to 6 cycles
  Arms: RO5083945 + cisplatin +gemcitabine
Drug: paclitaxel — up to 6 cycles
  Arms: RO5083945 + carboplatin + paclitaxel

SUMMARY:
This open-label, multicenter, non-randomized, dose-escalating phase Ib study with an expansion cohort will determine the recommended Phase II dose and schedule to investigate safety, tolerability, and activity of RO5083945 in combination with cisplatin and gemcitabine or carboplatin and paclitaxel in patients with advanced or recurrent non-small cell lung cancer of squamous histology who have not received prior chemotherapy for the metastatic disease. Cohorts of patients will receive escalating doses of RO5083945 in combination with up to 6 cycles of cisplatin and gemcitabine or carboplatin and paclitaxel. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Locally advanced (stage IIIB, excluding patients who are candidates for chemo-radiotherapy or radical thoracic radiotherapy), metastatic (stage IV) or recurrent squamous non-small cell lung cancer (NSCLC)
* Histologically documented squamous NSCLC. Mixed tumors should be categorized according to the predominant cell type
* Histological tumor tissue sample from initial diagnosis or new tumor biopsy representative of the disease
* Patients who have received adjuvant chemotherapy are eligible if the last administration of the prior adjuvant regimen occurred at least 3 months prior to enrollment
* At least one measurable disease lesion as per RECIST 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate hematological, liver and renal function
* Females of childbearing potential must commit to using a reliable and appropriate method of contraception until at least 3 months after the end of the last dose of study treatment

Exclusion Criteria:

* Prior chemotherapy (excluding neoadjuvant/adjuvant chemotherapy/chemo-radiotherapy) or treatment with another systemic anti-cancer agent (e.g. monoclonal antibody, tyrosine kinase inhibitor)
* Radiotherapy within the last 4 weeks prior to first dosing, except for limited field palliative radiotherapy for bone pain relief
* Treatment with any other investigational agent within 30 days prior to starting study treatment or participation in another clinical trial (e.g. CTC blood collection) within 7 days prior to starting study treatment
* Historical or clinical evidence of central nervous system (CNS) metastases (except for previously treated CNS metastases in patients that are asymptomatic, have had no evidence of active CNS metastases for >/= 3 months prior to first dose and have had no requirement for steroids or enzyme-inducing anticonvulsants in the last 14 days)
* Recent history of poorly controlled hypertension (systolic >180 mmHg or diastolic >100 mmHg)
* Severe uncontrolled illness, including poorly controlled diabetes mellitus and active or uncontrolled infection
* Hypersensitivity to the active substance or to any excipients or to any of the study drugs including premedication (corticosteroids, anti-histamine, paracetamol)
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose in combination with cisplatin and gemcitabine or carboplatin and paclitaxel | approximately 1.5 years
Recommended phase II dose (RP2D) of RO5083945 in combination with cisplatin and gemcitabine or carboplatin and paclitaxel | approximately 1.5 years

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 1.5 years
Pharmacokinetics: Serum concentrations of RO5083945 in combination with cisplatin and gemcitabine or carboplatin and paclitaxel | up to 18 weeks
Pharmacokinetics: Effect of RO5083945 on serum concentrations of cisplatin | up to 18 weeks
Pharmacokinetics: Effect of RO5083945 on serum concentrations of gemcitabine | up to 18 weeks
Pharmacokinetics: Effect of RO5083945 on serum concentrations of carboplatin | up to 18 weeks
Pharmacokinetics: Effect of RO5083945 on serum concentrations of paclitaxel | up to 18 weeks
Preliminary evidence of antitumor activity: Objective response rate (complete response, partial response and stable disease) | approximately 1.5 years
Duration of response | approximately 1.5 years
Biomarker assessments : Immune effector cells/EGFR markers | up to 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche